CLINICAL TRIAL: NCT05288634
Title: The Effect of Progressive Relaxation Exercise on Pain and Kinesiophobia After Lumbar Disc Herniation Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aksaray University (Other)
Responsible Party: Principal Investigator, Funda Cetinkaya, principal investigator, Aksaray University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2020/01-25
Record Dates: First submitted 2022-03-11; First posted 2022-03-21 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Lumbar Disc Herniation
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Routine maintenance and Progressive relaxation exercise practice
  Interventions: Other: Progressive relaxation exercise
- Control (No Intervention): Routine maintenance

INTERVENTIONS:
Other: Progressive relaxation exercise — Progressive relaxation exercise is a type of exercise that involves voluntary stretching and relaxation of major muscle groups in the human body, from the hands to the feet.
  Arms: Experimental

SUMMARY:
We aimed to assess the influence of progressive muscle relaxation exercise on kinesiophobia and pain during after lumbar disc surgery using the Visual Analog Scale (VAS) and the Tampa Kinesiophobia Scale in a prospective, randomized fashion.

DETAILED DESCRIPTION:
Lumbar disc herniation (LDH) is a common disease that is common in the society and limits the activities of individuals in daily life. Pain, which is an undesirable but expected result of surgical interventions, which are used in the treatment of diseases and play an important role in increasing the health level of people, is one of the most common postoperative complaints. The pain is sometimes severe enough to impede movement and causes paravertebral muscle spasm. Pain can also cause kinesiophobia, which is a factor that limits the person's physical activities. This study was conducted to determine the effect of progressive muscle relaxation exercises on kinesiophobia, which can be seen in parallel with pain in the postoperative period, on the pain level of patients after LDH surgery and on the kinesiophobia experienced in parallel.

The following hypotheses (H) were tested in this study:

H1. Progressive muscle relaxation exercise has an effect on reducing pain after LDH surgery.

H2. Progressive muscle relaxation exercise has an effect on reducing kinesiophobia after LDH surgery.

ELIGIBILITY:
Inclusion Criteria:

* • The patients included in the study had lumbar microdiscectomy surgery,

  * Patients aged 18 and over
  * Patients should not have any problems that would prevent them from expressing their pain level correctly and from understanding the information given,
  * The patients do not have any psychological disorders,
  * The patients do not have any other acute disease that will cause pain.

Exclusion Criteria:

* • Being diagnosed with a psychiatric disorder,

  * A complication (bleeding, hospital infection, etc.) developed in the patients before, during and after the operation within three days,
  * Not knowing Turkish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-12-29 (Actual)

PRIMARY OUTCOMES:
Tampa Kinesiophobia Scale | the day before the surgery
  : It is a 17-item scale. It gets a total score between 17-68. A high score on the scale indicates a high level of kinesiophobia.
Visual Analogue Scale | the day before the surgery
  It is the scale used to measure the severity of pain in patients. It is a scale whose beginning is -0- "no pain", and the other end is -10- "very severe pain" and each cm is given a numerical value at 1 centimeter (cm) intervals.

SECONDARY OUTCOMES:
Tampa Kinesiophobia Scale | third day after surgery
  It is a 17-item scale. It gets a total score between 17-68. A high score on the scale indicates a high level of kinesiophobia.
Visual Analogue Scale | third day after surgery
  It is the scale used to measure the severity of pain in patients. It is a scale whose beginning is -0- "no pain", and the other end is -10- "very severe pain" and each cm is given a numerical value at 1 centimeter (cm) intervals.

CONTACTS AND LOCATIONS:
Locations (1):
- Aksaray University, Aksaray, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No